CLINICAL TRIAL: NCT06884787
Title: Clinical and Subjective Evaluations of a Universal-Shade, Color Adjusting Resin Composite in Anterior Tooth Restorations: A Randomized Controlled Trial
Brief Title: Color Adjusting Resin Composite in Anterior Tooth Restorations: Clinical and Subjective Evaluations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20250094
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Composite Resins
Keywords: Single-sahde composite; Color adaptability,; Objective and subjective analysis; anterior restorations
MeSH Terms: interventions — Erythrocyte Count

STUDY DESIGN:
Intervention Model Description: Split mouth study design, patients will be assigned to two different treatment protocols.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor) The patients who participated in the study and the assessor of the treatment outcome do not know the type of treatment procedure received.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control group (Conventional RBC) (Experimental): Group 1 (n=120) teeth will be restored using conventional multi shade nanohybrid RBC (filtek Z350Xt,3M ESPE, San Paul, MN, USA)
  Interventions: Drug: Conventional nanohybrid multishade composite
- Test group (RBC with CAP) (Experimental): Group 2 (n=120) teeth will be restored using Omnichroma (single shade) composite with color adjustment postential (CAP). (Omnichroma, Tokuyama Dental, Tokio, Japan)
  Interventions: Drug: Single shade nanohybrid composite

INTERVENTIONS:
Drug: Conventional nanohybrid multishade composite — Teeth will be restored with conventional multi shade nanohybrid Resin Based Composite (RBC) filtek Z350Xt,3M ESPE, San Paul, MN, USA
  Other Names: Conventional resin based composite (RBC)
  Arms: Control group (Conventional RBC)
Drug: Single shade nanohybrid composite — Teeth will be restored with One-shade Resin Based Composite (Omnichroma, Tokuyama Dental, Tokio, Japan)
  Other Names: RBC with color adjustment potential (CAP)
  Arms: Test group (RBC with CAP)

SUMMARY:
The ability of single-shade composite restorations to blend with adjacent tooth structure shades is called chameleon effect. This effect is enhanced using specially designed spherical particles in the composite material which will help diffuse light in a way that mimics the natural color and translucency of teeth making the restoration nearly imperceptible to the naked eye.

The hypotheses of the investigation are as follow:

* Single-shade RBC exhibits similar shade matching and optical behavior to conventional RBC across all anterior restorations.
* Patient satisfaction regarding color blending between the restoration and tooth structure is comparable regardless of the type of material used.
* Dentist satisfaction regarding color blending is similar for both single-shade RBC and conventional RBC materials.

DETAILED DESCRIPTION:
Optimal shade matching in restorative dentistry is crucial for achieving aesthetic success, particularly in anterior restorations. This study aims to evaluate the shade-matching efficacy of single-shade resin-based composites (RBCs) in comparison to conventional multi-shade composite, using spectrophotometric analysis as an objective measurement tool. Additionally, the study assesses patient and clinician satisfactions with the color adaptability of single-shade composites across various restoration types, including Class V, III, IV, and diastema closures.

A sample of 240 teeth will be selected based on strict inclusion criteria and divided into two groups: a test group receiving single-shade RBCs and a control group receiving multi-shade composite. Each patient will receive at least one restoration from each treatment group, ensuring balanced comparison within subjects. Satisfaction levels regarding color adaptability and aesthetic integration will be evaluated using a Visual Analogue Scale (VAS) one-week post-treatment. The double-blind design will be employed as it maintains blinding for both patients and evaluating clinicians regarding the materials used in each restoration.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending the dental clinics at JUST in Irbid or on the university campus.
* Patients aged 18 years and older.
* Patients with good oral hygiene.
* Patients with a positive attitude towards dental treatment.
* Patients require restorations on at least two anterior teeth.
* Patients with spaces between teeth that do not require orthodontic treatment for correction.
* Patients with healthy pulp or reversible pulpitis.
* Patients without any periapical lesions

Exclusion Criteria:

* Teeth with enamel or dentin deformations.
* Teeth affected by fluorosis or tetracycline staining.
* Teeth with severe discoloration.
* Primary teeth.
* Patients with gingival inflammation or periodontal disease.
* Patients undergoing active orthodontic treatment.
* Heavy smokers.
* Very deep or very shallow cavities.
* Class IV cavities where more than half of the tooth surface is lost.
* Traumatic Class IV cavities with pulp exposure.
* Class III cavities that do not open labially.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Color measurements using digital spectrophotometer VITA Easyshade V. | 1 year
  The colour measurements will be taken at first session for each tooth in specific points as follow:
  1. One reading from middle part of tooth
  2. Three readings at three points around the restoration and 1 mm away from its margins.
  3. After one week and to give a chance for tooth rehydration and final color optimization a new reading will be obtained from the middle portion of the restoration.
  The color difference(∆E00) between the tooth structure around the restoration and the restoration itself will be calculated.
  The color difference(∆E00) between tooth and restoration will be compared between control and test group.
  The final ΔE00 value itself has no physical unit-it is just a numerical representation of color difference.
Subjective or Patient satisfaction | 1 year
  Patient satisfaction regarding the blending between the restoration and tooth surface will be recorded after one week using visual analogue scale (VAS).
  The scale is a horizontal line having 10 digits. Digit 0 starting from the right indicates total dissatisfaction regarding color blending between tooth and restoration and digit 10 indicates complete satisfaction.
  Patients will be asked to draw a line on VAS that represents their satisfaction regarding color matching and blending of the restoration.
  Measurements will be divided according following criteria:
  Poor: VAS values ranging from 0-5. Good :VAS values ranging from 5.1-10.
Objective or dentists satisfaction | 1 year
  Photographs of the restored teeth will be taken under standard setup using Canon 250DSLR camera, Sigma 105 mm Macro lens and Meike MK-14EXT TTL Macro Ring Flash.
  The pictures will be assessed by two calibrated dentists who did not know the restoration material being assessed. Blending with tooth surface will be done using VAS and the assessors will draw a line VAS.
  Measurements will be divided according following criteria:
  Poor: VAS values ranging from 0-5. Good :VAS values ranging from 5.1-10.

CONTACTS AND LOCATIONS:
Overall Officials: Zakereyya SM Albashaireh, Ph.D, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anwar RS, Hussein YF, Riad M. Optical behavior and marginal discoloration of a single shade resin composite with a chameleon effect: a randomized controlled clinical trial. BDJ Open. 2024 Feb 20;10(1):11. doi: 10.1038/s41405-024-00184-w. PMID 38378771
- [Background] Blum IR, Ozcan M. Reparative Dentistry: Possibilities and Limitations. Curr Oral Health Rep. 2018;5(4):264-269. doi: 10.1007/s40496-018-0191-1. Epub 2018 Sep 15. PMID 30524930
- [Background] Rashid F, Farook TH, Dudley J. Digital Shade Matching in Dentistry: A Systematic Review. Dent J (Basel). 2023 Oct 27;11(11):250. doi: 10.3390/dj11110250. PMID 37999014
- [Background] Barros MS, Silva PFD, Santana MLC, Braganca RMF, Faria-E-Silva AL. Background and surrounding colors affect the color blending of a single-shade composite. Braz Oral Res. 2023 Apr 28;37:e035. doi: 10.1590/1807-3107bor-2023.vol37.0035. eCollection 2023. PMID 37132724
- [Background] Leal CFC, Miranda SB, Alves Neto EL, Freitas K, de Sousa WV, Lins RBE, de Andrade AKM, Montes MAJR. Color Stability of Single-Shade Resin Composites in Direct Restorations: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Polymers (Basel). 2024 Jul 30;16(15):2172. doi: 10.3390/polym16152172. PMID 39125196
- [Background] Ahmed MA, Jouhar R, Khurshid Z. Smart Monochromatic Composite: A Literature Review. Int J Dent. 2022 Nov 8;2022:2445394. doi: 10.1155/2022/2445394. eCollection 2022. PMID 36398065
- [Background] Korkut B, Turkmen C. Longevity of direct diastema closure and recontouring restorations with resin composites in maxillary anterior teeth: A 4-year clinical evaluation. J Esthet Restor Dent. 2021 Jun;33(4):590-604. doi: 10.1111/jerd.12697. Epub 2020 Dec 23. PMID 33354867
- [Background] Cubukcu I, Gundogdu I, Gul P. Color match analysis of single-shade and multi-shade composite resins using spectrophotometric and visual methods after bleaching. Dent Mater J. 2023 Nov 29;42(6):826-834. doi: 10.4012/dmj.2023-115. Epub 2023 Oct 12. PMID 37821366
- [Background] Cruz da Silva ET, Charamba Leal CF, Miranda SB, Evangelista Santos M, Saeger Meireles S, Maciel de Andrade AK, Japiassu Resende Montes MA. Evaluation of Single-Shade Composite Resin Color Matching on Extracted Human Teeth. ScientificWorldJournal. 2023 Jun 26;2023:4376545. doi: 10.1155/2023/4376545. eCollection 2023. PMID 37404241
- [Background] Rohym S, Tawfeek HEM, Kamh R. Effect of coffee on color stability and surface roughness of newly introduced single shade resin composite materials. BMC Oral Health. 2023 Apr 22;23(1):236. doi: 10.1186/s12903-023-02942-y. PMID 37087507
- [Background] Zulekha, Vinay C, Uloopi KS, RojaRamya KS, Penmatsa C, Ramesh MV. Clinical performance of one shade universal composite resin and nanohybrid composite resin as full coronal esthetic restorations in primary maxillary incisors: A randomized controlled trial. J Indian Soc Pedod Prev Dent. 2022 Apr-Jun;40(2):159-164. doi: 10.4103/jisppd.jisppd_151_22. PMID 35859408
- [Background] Miranda AO, Favoreto MW, Matos TP, Castro AS, Kunz P, Souza JL, Carvalho P, Reis A, Loguercio AD. Color Match of a Universal-shade Composite Resin for Restoration of Non-carious Cervical Lesions: An Equivalence Randomized Clinical Trial. Oper Dent. 2024 Jan 1;49(1):20-33. doi: 10.2341/23-021-C. PMID 38057996